CLINICAL TRIAL: NCT05809505
Title: Feasibility and Safety of the 360-degree Turn Test Delivered Via Telehealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 360 Degree 1
Record Dates: First submitted 2023-03-09; First posted 2023-04-12 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
Keywords: telehealth; multiple sclerosis; 360-degree Turn Test
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The 360-degree turn test will be applied to patients first in the hospital environment and then by teleconference method, and the results will be recorded.
Masking Description: The researchers who evaluate the results and make statistics will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Sclerosis Patients (Experimental): Patients with a diagnosis of multiple sclerosis.
  Interventions: Diagnostic Test: 360-degree Turn Test; Other: Expanded Disability Status Scale; Other: Perceived Exertion

INTERVENTIONS:
Diagnostic Test: 360-degree Turn Test — The 360-degree turn test is a measure of dynamic balance. The person tested turns in a complete circle (360 degrees) while the time to complete and/or the number of steps to complete the turn is recorded.
Other: Expanded Disability Status Scale — The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with multiple sclerosis. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Other: Perceived Exertion — The Borg Rating of Perceived Exertion (RPE) is a way of measuring physical activity intensity level. Perceived exertion is how hard you feel like your body is working. It is based on the physical sensations a person experiences during physical activity, including increased heart rate, increased respiration or breathing rate, increased sweating, and muscle fatigue. Although this is a subjective measure, your exertion rating based on a 6 to 20 rating scale, may provide a fairly good estimate of your actual heart rate during physical activity.
  Other Names: Borg Scale

SUMMARY:
Walking, balance problems and falls are common in patients with multiple sclerosis. The 360-degree turn test is a test used to evaluate balance. Telerehabilitation is a rehabilitation system that has been increasingly used in recent years. Still, there is a need for studies on whether there is any difference between face-to-face evaluations with patients and telehealth methods. This study aims to investigate the feasibility and safety of the 360-degree turn test delivered via telehealth.

DETAILED DESCRIPTION:
The 360-degree turn test will be performed in the participant's home environment using a standardized protocol from previously published literature. Exercise professionals will administer the test during a single videoconferencing exercise appointment. Prior to the study commencement, clinicians will be given a 30-minute education session and written protocol to facilitate the standardized and safe performance of the test.

The test will be performed in the participant's home environment using videoconferencing. The clinician will explain the 360-degree turn test. Clinicians will record the device used by the participant. Where possible, participants will be instructed to adjust their device or camera to improve clinician visibility. The test will be stopped immediately if the participant reports increased pain, a moderate-significant increase in breathlessness, or is unsteady.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple sclerosis
* EDSS score ≤ 5.5

Exclusion Criteria:

* Not giving consent
* History of dislocation or surgery in the lower limbs
* History of fall within six months
* Any other disease, medication or intervention that can cause balance disturbance
* Patients who cannot use devices that is required for teleconference
* Patients that cannot understand English/ Turkish

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who safely completed the 360-degree turn test and completed the measurement in a way that could be used in clinical trials or follow-up | 1 day
  Feasibility and safety of the 360-degree turn test delivered via telehealth will be measured by the percived safety from researchers and results of the tests obtained from procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital
Locations (1):
- Başakşehir Çam ve Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request by the co-author.
Supporting Information: Study Protocol, SAP
Time Frame: One year
Access Criteria: Individual participant data will be shared upon reasonable request by the co-author.